CLINICAL TRIAL: NCT01090960
Title: An Open-Label, Phase I, Dose-Escalation Study Evaluating the Safety and Tolerability of GDC-0068 in Patients With Refractory Solid Tumors
Brief Title: A Study Evaluating the Safety and Tolerability of GDC-0068 in Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAM4743g; GO01335 (Other: Hoffmann-La Roche); 2009-015060-34 (EudraCT Number)
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Solid Cancers
MeSH Terms: interventions — ipatasertib

ARMS (1):
- A (Experimental)
  Interventions: Drug: GDC-0068

INTERVENTIONS:
Drug: GDC-0068 — Oral repeating dose

SUMMARY:
This is an open-label, multicenter, Phase I study to evaluate the safety, tolerability, and pharmacokinetics of escalating oral doses of GDC-0068 administered to patients with incurable, locally advanced or metastatic solid malignancy that has progressed or failed to respond to at least one prior regimen or for which there is no standard therapy. This study is expected to enroll approximately 39 to 57 patients at approximately two sites in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, incurable, locally advanced or metastatic solid tumors for which standard therapy either does not exist or has proven ineffective or intolerable.
* Evaluable or measurable disease
* Life expectancy >= 12 weeks
* Adequate hematologic and organ function within 14 days before initiation of GDC-0068
* Documented willingness to use an effective means of contraception (e.g., abstinence, hormonal or double barrier method, surgically sterilized partner) for both men and women while participating in the study

Exclusion Criteria:

* History of Type 1 or 2 diabetes mellitus requiring regular medication
* Grade > 2 hypercholesterolemia or hypertriglyceridemia
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Leptomeningeal disease as the only manifestation of the current malignancy
* Known untreated malignancies of the brain or spinal cord, or treated brain metastases that are not radiographically stable for >= 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events by NCI CTCAE grade and associated dose of GDC-0068 | Through study completion or early study discontinuation
Occurrence of dose-limiting toxicities (DLTs) by NCI CTCAE grade and associated dose of GDC-0068 | Through study completion or early study discontinuation
Occurrence of Grade 3 or 4 abnormalities in safety-related laboratory parameters and associated dose of GDC-0068 | Through study completion or early study discontinuation
PK parameters after single and multiple doses of GDC-0068 | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
Best overall response, duration of objective response, and progression-free survival (PFS) for patients with measurable disease according to RECIST | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Premal Patel, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (2):
- Spain (2):
  - Barcelona, Barcelona
  - Valencia, Valencia

REFERENCES:
- [Derived] Malhi V, Budha N, Sane R, Huang J, Liederer B, Meng R, Patel P, Deng Y, Cervantes A, Tabernero J, Musib L. Single- and multiple-dose pharmacokinetics, potential for CYP3A inhibition, and food effect in patients with cancer and healthy subjects receiving ipatasertib. Cancer Chemother Pharmacol. 2021 Dec;88(6):921-930. doi: 10.1007/s00280-021-04344-9. Epub 2021 Sep 1. PMID 34471960
- [Derived] Saura C, Roda D, Rosello S, Oliveira M, Macarulla T, Perez-Fidalgo JA, Morales-Barrera R, Sanchis-Garcia JM, Musib L, Budha N, Zhu J, Nannini M, Chan WY, Sanabria Bohorquez SM, Meng RD, Lin K, Yan Y, Patel P, Baselga J, Tabernero J, Cervantes A. A First-in-Human Phase I Study of the ATP-Competitive AKT Inhibitor Ipatasertib Demonstrates Robust and Safe Targeting of AKT in Patients with Solid Tumors. Cancer Discov. 2017 Jan;7(1):102-113. doi: 10.1158/2159-8290.CD-16-0512. Epub 2016 Nov 21. PMID 27872130
- [Derived] De Mattos-Arruda L, Weigelt B, Cortes J, Won HH, Ng CKY, Nuciforo P, Bidard FC, Aura C, Saura C, Peg V, Piscuoglio S, Oliveira M, Smolders Y, Patel P, Norton L, Tabernero J, Berger MF, Seoane J, Reis-Filho JS. Capturing intra-tumor genetic heterogeneity by de novo mutation profiling of circulating cell-free tumor DNA: a proof-of-principle. Ann Oncol. 2014 Sep;25(9):1729-1735. doi: 10.1093/annonc/mdu239. Epub 2014 Jul 9. PMID 25009010